CLINICAL TRIAL: NCT07350681
Title: Evaluation of the Effects of Orthognathic Surgery on Plantar Pressure Distribution and Posture
Brief Title: Effect of Orthognathic Surgery on Plantar Pressure and Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşenur Dindar (Other)
Responsible Party: Sponsor-Investigator, Ayşenur Dindar, Ayşenur Dindar, DDS, PhD in Orthodontics, Department of Orthodontics, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E.211678; 20240605E (Other Grant/Funding Number: Bezmialem Vakif University Scientific Research Projects Coordination Unit (BAP))
Record Dates: First submitted 2025-12-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Orthognathic Surgery; Postural Balance
MeSH Terms: interventions — Orthognathic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthognathic Surgery Group (Experimental): Patients undergoing orthognathic surgery with postoperative orthodontic treatment
  Interventions: Procedure: Orthognathic Surgery
- Control Group (No Intervention): Control group subjects not undergoing orthognathic surgery

INTERVENTIONS:
Procedure: Orthognathic Surgery — Participants in the experimental group will undergo orthognathic surgery
  Arms: Orthognathic Surgery Group

SUMMARY:
Orthognathic surgery leads to changes in the three-dimensional position of the jaws, which may result in alterations in head and neck posture as well as overall body posture. These postural changes are also expected to influence plantar pressure distribution. This study aims to evaluate the direction and magnitude of these changes by assessing posture and plantar pressure measurements before and after orthognathic surgery.

Postural analysis and plantar pressure measurements will be performed preoperatively and at the 6-month postoperative follow-up in patients undergoing orthognathic surgery. In order to allow a reliable comparison, a control group consisting of non-operated individuals will also be included. The range of natural changes observed in the control group will be determined, and the outcomes will be compared between the surgical and control groups.

By comparing preoperative and postoperative measurements, this study aims to evaluate the effects of orthognathic surgery on body posture and plantar pressure distribution. The findings are expected to contribute to the identification of parameters that should be considered in postoperative evaluation and rehabilitation. Furthermore, the results will provide valuable information regarding the postural and plantar pressure changes observed in patients following orthognathic surgery.

DETAILED DESCRIPTION:
A total of 60 participants will be included in the study, consisting of 30 patients scheduled to undergo orthognathic surgery as the study group and 30 patients who have completed their orthodontic treatment and attend regular follow-up visits as the control group.

In the study group, static and dynamic computerized plantar pressure analyses will be performed preoperatively using a pedobarography system (static analysis with BEVER®, dynamic analysis with PAROMED®). These analyses will be interpreted by a physiotherapist. Total body posture analysis will be performed using the PostureScreen® mobile application. Four-directional photographs of each participant will be taken by the researcher, and posture analysis will be conducted in collaboration with the physiotherapist according to the anatomical landmarks designated by the application. Body height and weight will be measured during routine pre-anesthetic evaluations. Preoperative lateral cephalometric radiographs (PLANMECA®) will be obtained as part of routine clinical records, and cephalometric evaluations will be performed on these images.

At the 6-month postoperative follow-up, body height and weight measurements, lateral cephalometric radiographs, static and dynamic computerized plantar pressure analyses, and total body posture analysis will be repeated in the surgical group. Baseline and follow-up values will be compared to determine the direction and magnitude of changes.

In the control group, in addition to routine lateral cephalometric radiographs obtained at the end of treatment, total body posture analysis using the PostureScreen® mobile application, static and dynamic computerized plantar pressure analyses, and body height and weight measurements will be performed. The same assessments will be repeated at the routine 6-month follow-up visit for the control group participants.

ELIGIBILITY:
Inclusion Criteria:

* Study Group (Orthognathic Surgery Group)

Participants will be eligible for inclusion in the surgical cohort if they meet all of the following criteria:

Individuals scheduled to undergo single-jaw or double-jaw orthognathic surgery as part of comprehensive orthodontic treatment.

Currently receiving orthodontic therapy utilizing clear aligner systems or fixed orthodontic appliances.

Availability of preoperative lateral cephalometric radiographs obtained as part of routine clinical evaluation.

Age ≥ 18 years at the time of enrollment.

Completion of a minimum of 6 months of postoperative orthodontic treatment, enabling standardized follow-up evaluation.

Body Mass Index (BMI) < 30 kg/m², to minimize confounding effects related to obesity on postural and plantar pressure measurements.

Control Group (Non-surgical Group)

Participants will be eligible for inclusion in the control cohort if they meet all of the following criteria:

Individuals not undergoing orthognathic surgery during the study period.

Receiving orthodontic treatment with clear aligners or fixed appliances, comparable to the surgical cohort.

BMI < 30 kg/m².

Age ≥ 18 years.

No participation in physical activities or rehabilitative programs that may alter postural parameters or plantar pressure distribution during the study period.

Exclusion Criteria:

* Participants from either cohort will be excluded if they exhibit:

Neuromuscular, musculoskeletal, or postural disorders that may independently influence balance or plantar pressure distribution.

History of previous orthognathic or maxillofacial surgery.

Systemic diseases affecting bone metabolism, neuromuscular function, or gait.

Pregnancy.

Inability or unwillingness to comply with study procedures or follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Plantar Pressure Distribution | Baseline and 6 months postoperative
  Plantar pressure distribution will be evaluated using static and dynamic pedobarographic measurements. Peak plantar pressure, pressure distribution patterns, and contact area will be recorded preoperatively and at 6 months postoperatively to assess changes in plantar loading following orthognathic surgery.

SECONDARY OUTCOMES:
Change in Whole-Body Postural Alignment Measured by PostureScreen® Mobile Application at Baseline and 6 Months Postoperative | Preoperative baseline and 6 months postoperative
  Whole-body postural alignment will be quantitatively evaluated using the PostureScreen® mobile application. Digital postural parameters will be recorded preoperatively and at 6 months postoperatively to assess changes in global body posture following orthognathic surgery.
Change in Cranio-Cervical Posture Measured by Lateral Cephalometric Analysis at Baseline and 6 Months Postoperative | Baseline & 6 months postoperative
  Cranio-cervical posture will be assessed using lateral cephalometric radiographs. Angular cephalometric parameters will be recorded preoperatively. OPT/CVT angle (Odontoid Process Tangent / Cervical Vertebra Tangent angle) will be measured on lateral cephalometric radiographs to evaluate postoperative cranio-cervical postural changes.

CONTACTS AND LOCATIONS:
Overall Officials: AYSENUR DİNDAR, Principal Investigator — Bezmiâlem Vakıf University, Institute of Health Sciences, Department of Orthodontics, İstanbul, Türkiye
Locations (1):
- Bezmialem Vakif University Faculty of Dentistry, Department of Orthodontics, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No